CLINICAL TRIAL: NCT01322126
Title: Comparison of Safety And Efficacy of Neyraxial Anesthesia,Palpation Versus Ultrasound
Brief Title: Comparison of Safety And Efficacy of Neuraxial Anesthesia, Palpation Versus Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Saifi Fayez, Hadassah Medical Organization, Israel Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00710-HMO-CTIL
Record Dates: First submitted 2011-03-07; First posted 2011-03-24 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-03

CONDITIONS: Regional Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ultrasound ,without ultrasound (Experimental): ultrasound group will be passed the neuraxial anesthesia with ultrasound,the secoud group will be passed the neuraxial anesthesia without ultrasound .
  Interventions: Device: ultrasound probe

INTERVENTIONS:
Device: ultrasound probe — we will compare two technique of neuraxial anesthesia;one group will be passed neuraxial anesthesia with the intervention the ultrasound and the other group without the intervention of the ultrasound.

SUMMARY:
The purpose of this study is to determine whether use of the ultrasound to locate the epidural space and assist with performing neuraxial anesthesia will decrease numbers of the attempts required for successful placement of epidural catheter.

DETAILED DESCRIPTION:
It is known that ultrasound can be useful to assist placement of epidural analgesia among pregnant women.extenseve research on the usefulness of ultrasound imaging to facilitate the placement of neuraxial anesthesia in pregnant have been done.The potential advantages of successful placement among non-pregnant patients include increases the safety and comfort.

In our study all patients schedueld to receive an nueraxial anesthesia for non-obstetric surgery will be included.The investigator will request permission from the Helsinki committee of hadassah university hospital.Patients will be requesting for surgery and will be randomized to one of two study groups.One group will be passed neuraxial anesthesia on the standart technique and the secound group will be passed neuraxial anesthesia with the help of ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for neuraxial anesthesia

Exclusion Criteria:

* previous spine surgery
* contraindication for neuraxial anesthesia
* refusing to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Number of epidural attempts made to succeed for placing epidural needle and catheter in epidural space | one year
  Each attempt at placing epidural needle in epidural space will be recorded. Total number of attempts will be recorded

SECONDARY OUTCOMES:
patient satisfaction as measured by VAS (0=not satisfied, 10 = most satisfied) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fayez T Saifi, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel